CLINICAL TRIAL: NCT00681174
Title: Preoperative Controlled-Release Oxycodone or Intraoperative Morphine As Transition Opioid After Intravenous Anesthesia For Video-Assisted Thoracic Surgery: a Randomized, Double-blind, Controlled Trial.
Brief Title: Controlled-Release Oxycodone For Postoperative Analgesia After Video-Assisted Thoracic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to enroll sufficient patients by expected deadline.
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Guido Fanelli, Professor of Anesthesiology and Critical Care Medicine, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANEST-TOR-01
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Anesthesia Recovery Period; Pain, Postoperative
Keywords: Care, Postoperative; Analgesia; Analgesics, Opioid; Morphine; Remifentanil; Oxycodone; Anesthesia, Regional; Anesthesia, Intravenous; Preanesthetic Medication; Analgesia, Patient-Controlled
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Morphine; Oxycodone; Ropivacaine; Propofol; Remifentanil; Acetaminophen; Passive Cutaneous Anaphylaxis; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Control intervention will be intraoperative i.v. morphine administration 30 minutes before the end of anesthesia.
  Interventions: Drug: Morphine; Procedure: Paravertebral block; Drug: Propofol; Drug: Remifentanil; Drug: Paracetamol
- CROxy (Experimental): The intervention group will receive controlled-release oxycodone 1 h pre-operatively
  Interventions: Drug: oxycodone; Procedure: Paravertebral block; Drug: Propofol; Drug: Remifentanil; Drug: Paracetamol; Drug: Morphine

INTERVENTIONS:
Drug: Morphine — 0.15 mg/kg i.v. bolus, 30 minutes before the expected end of anesthesia
  Arms: Control
Drug: oxycodone — 20 mg p.o. 1 h before the start of anesthesia
  Other Names: controlled-release oxycodone; CR oxycodone; OxyContin®
  Arms: CROxy
Procedure: Paravertebral block — * Three injections of 0.5% ropivacaine, 5 ml each
  * Injections at the T5, T6 and T7 levels
  A 22G spinal needle will be used to contact the ipsilateral transverse process; the needle will be "walked off" the process and the injection will be made 1 cm deeper.
  Other Names: Paravertebral nerve block; Naropin®
Drug: Propofol — * Plasma concentration target-controlled infusion based on bispectral index values
  * Acceptable range of concentrations: 2-4 µg/mL
  * Target bispectral index values: 40-60
  * Infusion starts at 4 µg/ml target, after pre-oxygenation (i.e., start of anesthesia)
  Other Names: Propofol TCI; target-controlled infusion; TIVA; TCI-TIVA; TIVA-TCI; Diprivan®
Drug: Remifentanil — * 50 µg/mL i.v. solution infused at 0.05-0.2 µg/kg/min
  * Infusion starts 7 min before propofol infusion (i.e., start of anesthesia)
  * Infusion rate adjusted to maintain mean arterial blood pressure within ±20% of baseline values.
  * Infusion stopped after end of surgery and after patients are brought back to the supine position (i.e., end of anesthesia)
  Other Names: TIVA; Ultiva®
Drug: Paracetamol — 1 g i.v. bolus 30 min before the end of anesthesia; 1 g i.v. bolus q8h thereafter.
  Other Names: Acetaminophen; Perfalgan®
Drug: Morphine — Patient-controlled intravenous infusion pump (IV-PCA).
  * 50 mg morphine in 50 ml saline solution (1 mg/ml)
  * Incremental dose: 1 mg
  * Lock-out time: 8 min
  * Limit: 40 mg in 4 h
  * Background infusion: none
  Other Names: PCA; IVPCA; IV-PCA; PCA-IV; Patient-controlled analgesia

SUMMARY:
The main hypothesis of this study is that preoperative administration of controlled-release (CR) oxycodone may reduce acute postoperative pain and improve time to discharge from the post-anesthesia care unit in patients undergoing video-assisted thoracoscopy for spontaneous pneumothorax.

The study drug will be compared with intravenous morphine administered 30 minutes before the end of anesthesia.

DETAILED DESCRIPTION:
Although spontaneous pneumothorax may be treated conservatively by simple observation or chest tube insertion, up to 50% of patients treated conservatively may experience recurrence in subsequent months or years.

Video-assisted thoracic surgery (VATS) is a minimally-invasive surgical approach to treat spontaneous pneumothorax and reduce the risk of recurrence. Compared to open thoracotomy, VATS may facilitate a faster recovery and lead to earlier home discharge.

Totally-intravenous anesthesia (TIVA) with propofol and remifentanil is a useful anesthetic technique for VATS, as the drugs are rapidly eliminated after the end of the procedure, leading to fast recovery from anesthesia.

One drawback of ultra-short-acting opioid remifentanil is residual hyperalgesia after the end of the infusion, particularly after VATS, which is associated with relatively short but intense pain after surgery.

Intravenous morphine, administered just before the end of anesthesia, is the typical choice for pain relief after TIVA. However, this drug may require repeated titration and may be associated with postoperative nausea and vomiting, itchiness or drowsiness in the early postoperative period.

Oxycodone, another opioid, is available in an oral controlled-release (CR) formulation which grants relatively constant plasma levels of the drug after 1 h of administration.

The investigators hypothesize that administration of CR oxycodone 20 mg 1 hour before surgery may lead to better recovery parameters in the post-anesthesia care unit, thus granting earlier discharge to the surgical ward.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for video-assisted thoracic surgery for clinical diagnosis of spontaneous pneumothorax
* Must be able to swallow tablets 1 h before surgery
* American Society of Anesthesiologists (ASA) physical status class I or II

Exclusion Criteria:

* Known allergy or other contraindications to study drugs
* Acute myocardial infarction ≤6 months before enrollment
* Serum creatinine > 2 mg/dL
* Body mass index (BMI) > 30
* Diagnosis of psychiatric disorders
* Known or possible pregnancy
* Epilepsy
* Chronic opioid therapy or abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Morphine consumption (intravenous titration in PACU + i.v. patient-controlled pump usage) | 48 h

SECONDARY OUTCOMES:
Pain intensity as measured on a visual analog scale | 1 h after end of anesthesia
Time to discharge from post-anesthesia care unit (Aldrete score >9) | 0-12 h after end of anesthesia
Nausea or vomiting | 48 h
Respiratory depression (SpO2 < 92% or respiratory rate <8) | 48 h

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — Section of Anesthesiology and Critical Care, Dept. of Anesthesiology, University of Parma, Italy; Marco Berti, MD, Study Director — II Unit of Anesthesia, Critical Care and Pain Medicine, University Hospital of Parma, Italy; Franca Bridelli, MD, Principal Investigator — II Unit of Anesthesia, Critical Care and Pain Medicine, University Hospital of Parma, Italy
Locations (1):
- University Hospital / Azienda Ospedaliero-Universitaria, Parma, PR, Italy

REFERENCES:
- [Background] Noppen M, Baumann MH. Pathogenesis and treatment of primary spontaneous pneumothorax: an overview. Respiration. 2003 Jul-Aug;70(4):431-8. doi: 10.1159/000072911. PMID 14512683
- [Background] Hansen EG, Duedahl TH, Romsing J, Hilsted KL, Dahl JB. Intra-operative remifentanil might influence pain levels in the immediate post-operative period after major abdominal surgery. Acta Anaesthesiol Scand. 2005 Nov;49(10):1464-70. doi: 10.1111/j.1399-6576.2005.00861.x. PMID 16223391
- [Background] Sunshine A, Olson NZ, Colon A, Rivera J, Kaiko RF, Fitzmartin RD, Reder RF, Goldenheim PD. Analgesic efficacy of controlled-release oxycodone in postoperative pain. J Clin Pharmacol. 1996 Jul;36(7):595-603. doi: 10.1002/j.1552-4604.1996.tb04223.x. PMID 8844441
- [Background] Vogt A, Stieger DS, Theurillat C, Curatolo M. Single-injection thoracic paravertebral block for postoperative pain treatment after thoracoscopic surgery. Br J Anaesth. 2005 Dec;95(6):816-21. doi: 10.1093/bja/aei250. Epub 2005 Sep 30. PMID 16199417
- [Background] Kaya FN, Turker G, Basagan-Mogol E, Goren S, Bayram S, Gebitekin C. Preoperative multiple-injection thoracic paravertebral blocks reduce postoperative pain and analgesic requirements after video-assisted thoracic surgery. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):639-43. doi: 10.1053/j.jvca.2006.03.022. Epub 2006 Aug 8. PMID 17023279